CLINICAL TRIAL: NCT00028639
Title: A Phase II Study of the Proteasome Inhibitor PS-341 (NSC 681 239) in Patients With Metastatic Breast Cancer
Brief Title: PS-341 in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: William Gradishar, MD, Northwestern University
Purpose: Treatment
Other Study IDs: NCI 00B11; NU-NCI00B11; NCI-1862
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
RATIONALE: PS-341 may stop the growth of tumor cells by blocking the enzymes necessary for cancer cell growth.

PURPOSE: Phase II trial to study the effectiveness of PS-341 in treating women who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective tumor response in women with metastatic breast cancer treated with bortezomib.
* Determine the toxic effects of this drug in these patients.
* Determine the progression-free survival in patients treated with this drug.

OUTLINE: Patients receive bortezomib IV over 3-5 seconds twice weekly for 2 weeks. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 12-35 patients will be accrued for this study within 6-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Metastatic disease
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR
  * At least 10 mm by spiral CT scan
* Previously treated with 1 prior chemotherapy regimen (with or without trastuzumab [Herceptin]) for metastatic disease

  * Relapse during or within 6 months after completion of adjuvant chemotherapy considered treatment failure
* No known brain metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* SGOT/SGPT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other:

* No uncontrolled concurrent illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to bortezomib
* No other prior malignancy within the past 5 years unless curatively treated and disease free
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy:

* Prior hormonal therapy for metastatic disease allowed
* At least 4 weeks since prior hormonal therapy and recovered

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* Prior adjuvant therapy allowed
* At least 4 weeks since prior investigational drugs and recovered
* No other concurrent investigational or commercial agents or therapies for breast cancer
* No concurrent combination antiretroviral therapy for HIV

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-08; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J. Gradishar, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States